CLINICAL TRIAL: NCT01440374
Title: A Three-part Study of Eltrombopag in Thrombocytopenic Subjects With Myelodysplastic Syndromes or Acute Myeloid Leukemia (Part 1: Open-label, Part 2: Randomized, Double-blind, Part 3: Extension)
Brief Title: A Three-part Study of Eltrombopag in Thrombocytopenic Subjects With Myelodysplastic Syndromes or Acute Myeloid Leukemia
Acronym: ASPIRE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 114968; 2011-000114-19 (EudraCT Number)
Record Dates: First submitted 2011-09-15; First posted 2011-09-26 (Estimated); Results first posted 2016-06-14 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-05

CONDITIONS: Thrombocytopaenia
Keywords: acute myeloid leukemia (AML); acute myelogenous leukemia (AML); acute non lymphocytic leukemia (ANLL); myeloproliferative disease (MDS); myelodysplastic syndrome ( secondary acute myeloid leukemia); refractory acute myeloid leukemia
MeSH Terms: conditions — Thrombocytopenia; Leukemia, Myeloid, Acute; Myeloproliferative Disorders; Myelodysplastic Syndromes | interventions — eltrombopag

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Part 1, Open Label (Experimental): 100 mg daily (50 mg for subjects of East Asian heritage), intrasubject dose escalations to a maximum dose 300 mg (150 mg for subjects of East Asian heritage) are allowed.
  Interventions: Drug: eltrombopag
- Part 2, eltrombopag arm (Experimental): 100 mg daily (50 mg for subjects of East Asian heritage), intra-subject dose escalations to a maximum dose of 300 mg (150 mg for subjects of East Asian heritage)
  Interventions: Drug: eltrombopag
- Part 2, placebo arm (Experimental): 100 mg matching placebo daily (50 mg for subjects of East Asian heritage), intra-subject dose escalations to a maximum dose of 300 mg matching placebo (150 mg for subjects of East Asian heritage)
  Interventions: Drug: placebo
- part 3 extension (Experimental): 100 mg daily (50 mg for subjects of East Asian heritage), intra-subject dose escalations to a maximum dose of 300 mg (150 mg for subjects of East Asian heritage)
  Interventions: Drug: eltrombopag

INTERVENTIONS:
Drug: eltrombopag — 100 mg daily (50 mg for subjects of East Asian heritage), intra-subject dose escalations to a maximum dose of 300 mg (150 mg for subjects of East Asian heritage)
  Other Names: Promacta
  Arms: Part 1, Open Label; Part 2, eltrombopag arm; part 3 extension
Drug: placebo — 100 mg matching placebo daily (50 mg for subjects of East Asian heritage), intra-subject dose escalations to a maximum dose of 300 mg matching placebo (150 mg for subjects of East Asian heritage)
  Arms: Part 2, placebo arm

SUMMARY:
This was a worldwide, three-part (Part 1: open-label, Part 2: randomized, double-blind, Part 3: extension), multi-center study to evaluate the effect of eltrombopag in subjects with myelodysplastic syndromes (MDS) or acute myeloid leukemia (AML) who have thrombocytopenia due to bone marrow insufficiency from their underlying disease or prior chemotherapy. This objective was assessed by a composite primary endpoint that consists of the following: the proportion of ≥Grade 3 hemorrhagic adverse events, or platelet counts <10 Gi/L, or platelet transfusions. Patients with MDS or AML and Grade 4 thrombocytopenia due to bone marrow insufficiency from their underlying disease or prior chemotherapy were enrolled in the study. No low or intermediate-1 risk MDS subjects were enrolled in the study. Subjects must have had at least one of the following during the 4 weeks prior to enrolment: platelet count <10 Gi/L, platelet transfusion, or symptomatic hemorrhagic event. Supportive standard of care (SOC), including hydroxyurea, was allowed as indicated by local practice throughout the study. The study had 3 sequential parts. Subjects who were enrolled in Part 1 (open-label) cannot be enrolled in Part 2 of the study (randomized, double-blind); however, subjects who completed the treatment period for Part 1 or Part 2 (8 and 12 weeks, respectively) continued in Part 3 (extension) if the investigator determined that the subject was receiving clinical benefit on treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (18 years of age or older) with MDS or AML (bone marrow blasts ≤50%) with thrombocytopenia due to bone marrow insufficiency from the disease or prior treatment. Subjects with transient thrombocytopenia due to active treatment with disease modifying agents or chemotherapy (except for hydroxyurea) are excluded.
* Subjects must have Grade 4 thrombocytopenia (platelet counts <25 Gi/L) due to bone marrow insufficiency (or Grade 4 thrombocytopenia, but platelet count greater than or equal to 25 Gi/L due to platelet transfusion). In addition, subjects must have had at least one of the following during the 4 week screening period: platelet transfusion, or symptomatic bleeding or platelet count <10 Gi/L. Subjects whose thrombocytopenia below 10 Gi/L is due to causes other than bone marrow insufficiency (e.g., fever, infection, autoimmune disease) are not eligible.
* Subjects must have platelet count, bleeding and platelet transfusion data available over a period of at least 4 weeks prior to randomization.
* Prior systemic treatment for malignancy, with the exception of hydroxyurea, must have been discontinued prior to entry into the study: at least 4 weeks before Day 1 for the following: chemotherapy, demethylating agents (azacitidine or decitabine), lenalidomide, thalidomide, clofarabine and IL-11(oprelvekin); at least 8 weeks before Day 1 for antithymocyte/antilymphocyte globulin.
* Subjects with a prior stem cell transplant (SCT) must have relapsed after the SCT.
* Subjects must be stable and, in the opinion of the investigator, be expected to complete a 12 week treatment period.
* ECOG Status 0-2.
* Subject must be able to understand and comply with protocol requirements and instructions.
* Subject has signed and dated an informed consent form.
* Adequate baseline organ function defined by the criteria below: total bilirubin ≤ 1.5xULN except for Gilbert's syndrome or cases clearly not indicative of inadequate liver function (i.e. elevation of indirect (hemolytic) bilirubin in the absence of ALT abnormality), ALT ≤ 3xULN, creatinine ≤ 2.5xULN
* Women must be either of non-child bearing potential or women with child-bearing potential and men with reproductive potential must be willing to practice acceptable methods of birth control during the study Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to the first dose of study treatment.
* In France, a subject eligible for inclusion in this study only if either affiliated to, or a beneficiary of, a social security category.

Exclusion Criteria:

* Subjects with MDS and an IPSS of low or intermediate-1 risk at screening.
* Subjects with a diagnosis of acute promyelocytic or megakaryocytic leukemia or AML secondary to a myeloproliferative neoplasm.
* History of treatment with romiplostim or other TPO-R agonists.
* Subjects with a QTc >480 msec (QTc >510 msec for subjects with Bundle Branch Block).
* Leukocytosis ≥25,000/uL on Day 1 of treatment with study medication.
* Subjects with known thrombophilic risk factors. Exception: Subjects for whom the potential benefits of participating in the study outweigh the potential risks of thromboembolic events, as determined by the investigator.
* Female subjects who are nursing or pregnant (positive serum or urine β-human chorionic gonadotropin [β-hCG] pregnancy test) at screening or pre-dose on Day 1.
* Current alcohol or drug abuse.
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication.
* Active and uncontrolled infections (e.g. sepsis, hepatitis B, hepatitis C).
* Subjects infected with Human Immunodeficiency Virus (HIV).
* Subjects with liver cirrhosis (as determined by the investigator).
* Subjects receiving or planned to receive any prohibited medication.
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to eltrombopag or excipient (microcrystalline cellulose, mannitol, polyvinylpyrrolidone, sodium starch glycolate, magnesium stearate, hypromellose, titanium dioxide, polyethylene glycol 400 and polysorbate 80) that contraindicates the subjects' participation.
* In France, subjects who have participated in any study using an investigational drug during the previous 30 days.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2011-09; Primary Completion 2015-03 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (111):
- United States (18):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Hot Springs, Arkansas
  - Novartis Investigative Site, Jonesboro, Arkansas
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Stanford, California
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, West Palm Beach, Florida
  - Novartis Investigative Site, Augusta, Georgia
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Kansas City, Missouri
  - Novartis Investigative Site, Hackensack, New Jersey
  - Novartis Investigative Site, Voorhees Township, New Jersey
  - Novartis Investigative Site, The Bronx, New York
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Milwaukee, Wisconsin
- Argentina (4):
  - Novartis Investigative Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Novartis Investigative Site, La Plata, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Ciudad AutÃ³noma de Buenos Aires
- Belgium (7):
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Brasschaat
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Yvoir
- Brazil (10):
  - Novartis Investigative Site, Goiânia - GO, Goiás
  - Novartis Investigative Site, GoiÃ¢nia - GO, GoiÃ¡s
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Curitiba, ParanÃ¡
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Barretos, São Paulo
  - Novartis Investigative Site, Barretos, SÃ£o Paulo
  - Novartis Investigative Site, SÃ£o Paulo, SÃ£o Paulo
  - Novartis Investigative Site, Rio de Janeiro
  - Novartis Investigative Site, São Paulo
- Canada (3):
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Czechia (2):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Prague
- Germany (6):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Stuttgart, Baden-Wurttemberg
  - Novartis Investigative Site, Göttingen, Lower Saxony
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Düsseldorf, North Rhine-Westphalia
  - Novartis Investigative Site, Dresden, Saxony
- Greece (4):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Heraklion, Crete
  - Novartis Investigative Site, Ioannina
  - Novartis Investigative Site, Thessaloniki
- Hong Kong (2):
  - Novartis Investigative Site, Chai Wan
  - Novartis Investigative Site, Shatin, New Territories
- Hungary (5):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Kaposvár
  - Novartis Investigative Site, KaposvÃ¡r
  - Novartis Investigative Site, Szeged
- Ireland (6):
  - Novartis Investigative Site, Cork
  - Novartis Investigative Site, Dublin
  - Novartis Investigative Site, James Street
  - Novartis Investigative Site, Limerick
  - Novartis Investigative Site, Tallaght, Dublin
  - Novartis Investigative Site, Tullamore
- Israel (8):
  - Novartis Investigative Site, Beersheba
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Holon
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Rehovot
  - Novartis Investigative Site, Tel Aviv
- Italy (5):
  - Novartis Investigative Site, Bologna, Emilia-Romagna
  - Novartis Investigative Site, Brescia, Lombardy
  - Novartis Investigative Site, Milan, Lombardy
  - Novartis Investigative Site, Alessandria, Piedmont
  - Novartis Investigative Site, Florence, Tuscany
- Mexico (5):
  - Novartis Investigative Site, Monterrey, Nuevo LeÃ³n
  - Novartis Investigative Site, Monterrey, Nuevo León
  - Novartis Investigative Site, Chihuahua City
  - Novartis Investigative Site, Mexico City
  - Novartis Investigative Site, Oaxaca City
- Novartis Investigative Site, Amsterdam, Netherlands
- Poland (3):
  - Novartis Investigative Site, Chorzów
  - Novartis Investigative Site, Torun
  - Novartis Investigative Site, Warsaw
- Novartis Investigative Site, San Juan, Puerto Rico
- Russia (4):
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Petrozavodsk
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, St'Petersburg
- South Korea (2):
  - Novartis Investigative Site, Hwasun
  - Novartis Investigative Site, Seoul
- Spain (9):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Granada
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, MÃ¡laga
  - Novartis Investigative Site, Pozuelo de AlarcÃ³n/Madrid
  - Novartis Investigative Site, Pozuelo de Alarcón/Madrid
  - Novartis Investigative Site, Salamanca
  - Novartis Investigative Site, Santander
- Taiwan (3):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Tainan County
  - Novartis Investigative Site, Taoyuan
- Thailand (3):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Khon Kaen
  - Novartis Investigative Site, Songkhla

REFERENCES:
- [Derived] Mittelman M, Platzbecker U, Grosicki S, Lawniczek T, Zhu Z, Selleslag D. Long-Term Safety and Efficacy of Eltrombopag for Advanced Myelodysplastic Syndromes or Acute Myeloid Leukemia and Severe Thrombocytopenia: Results of the ASPIRE Extension Study. Acta Haematol. 2023;146(5):373-378. doi: 10.1159/000531146. Epub 2023 May 19. PMID 37231838
- [Derived] Mittelman M, Platzbecker U, Afanasyev B, Grosicki S, Wong RSM, Anagnostopoulos A, Brenner B, Denzlinger C, Rossi G, Nagler A, Garcia-Delgado R, Portella MSO, Zhu Z, Selleslag D. Eltrombopag for advanced myelodysplastic syndromes or acute myeloid leukaemia and severe thrombocytopenia (ASPIRE): a randomised, placebo-controlled, phase 2 trial. Lancet Haematol. 2018 Jan;5(1):e34-e43. doi: 10.1016/S2352-3026(17)30228-4. Epub 2017 Dec 11. PMID 29241762

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part 1, 17 subjects received open-label eltrombopag. Part 2, 145 subjects were randomized to receive eltrombopag plus SOC (N=98) or placebo plus SOC (N=47).
  Part 3, 59 subjects from Part 2 entered Part 3. SOC was allowed as needed throughout the study. Subjects could receive disease-modifying therapy as needed.
Pre-assignment Details: Participants with myelodysplastic syndromes (MDS) or acute myeloid leukemia (AML) and Grade 4 thrombocytopenia due to bone marrow insufficiency and had at least one of the following: platelet count <10 Giga cells per liter, platelet transfusion or symptomatic hemorrhagic event during the 4 weeks prior to enrollment, were enrolled in the study.
Groups:
- Part 1: Eltrombopag: The eltrombopag starting dose the participants received was 100 milligrams (mg) daily (50 mg for participants of East Asian heritage). The dose of eltrombopag was escalated from 100 mg to 200 mg (50 mg to 100 mg for East Asians) and further from 200 mg to 300 mg once daily (100 mg to 150 mg for East Asians) based on the platelet response and safety data after two weeks of current dose level. After all participants finished the 8 week treatment period, platelet response and safety were analyzed before initiating Part 2 of the study. Supportive standard of care was allowed as needed. The duration of Part 1 was 8 weeks.
- Part 2: Placebo: Participants received eltrombopag matching placebo once daily (3 tablets). Supportive standard of care was allowed as needed throughout the study.
- Part 2: Eltrombopag: The eltrombopag starting dose the participants received was 100 mg daily (50 mg for participants of East Asian heritage). The duration of treatment with the initial dose level prior to first dose escalation was determined based on the platelet response and toxicity observed in Part 1. The dose of eltrombopag was escalated from 100 mg to 200 mg (50 mg to 100 mg for East Asians) and further from 200 mg to 300 mg once daily (100 mg to 150 mg for East Asians) based on the platelet response and safety data after two weeks of current dose level. Supportive standard of care was allowed as needed throughout the study.
- Part 3: Eltrombopag: 23 subjects of the 47 randomized to the placebo group in Part 2 entered part 3. 36 subjects of the 98 randomized to the Etrombopag group in Part 2 entered part 3.
  All subjects received eltrombopag. Part 3 subjects could also have received treatment for their disease per local SOC, including azacitidine, decitabine, lenalidomide, and chemotherapy. The duration of Part 3 was to be 10 months for subjects from Part 1and 9 months for subjects from Part 2.
Period: Part 1: Open-label Phase
Arm/Group | Part 1: Eltrombopag | Part 2: Placebo | Part 2: Eltrombopag | Part 3: Eltrombopag
Started | 17 | 0 | 0 | 0
Completed | 11 | 0 | 0 | 0
Not Completed | 6 | 0 | 0 | 0
Not completed — Adverse Event | 5 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Period: Part 2; Double-blind Phase
Arm/Group | Part 1: Eltrombopag | Part 2: Placebo | Part 2: Eltrombopag | Part 3: Eltrombopag
Started | 0 | 47 | 98 | 0
Completed | 0 | 27 | 43 | 0
Not Completed | 0 | 20 | 55 | 0
Not completed — Physician Decision | 0 | 8 | 17 | 0
Not completed — Withdrawal by Subject | 0 | 4 | 5 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 7 | 31 | 0
Not completed — Not treated | 0 | 0 | 1 | 0
Period: Part 3: Extension
Arm/Group | Part 1: Eltrombopag | Part 2: Placebo | Part 2: Eltrombopag | Part 3: Eltrombopag
Started | 0 | 0 | 0 | 59
Completed | 0 | 0 | 0 | 27
Not Completed | 0 | 0 | 0 | 32
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 13
Not completed — Physician Decision | 0 | 0 | 0 | 14

BASELINE CHARACTERISTICS:
Population: Part 3, 59 subjects from Part 2 entered Part 3 (23 of 47 subjects in the placebo group in Part 2 and 36 of 98 subjects in the eltrombopag group in Part 2). All subjects who entered Part 3 received treatment with eltrombopag. SOC was allowed as needed throughout the study. Subjects could receive disease-modifying therapy as needed.
Groups:
- Part 1: Eltrombopag: The eltrombopag starting dose the participants received was 100 mg daily (50 mg for participants of East Asian heritage). The dose of eltrombopag was escalated from 100 mg to 200 mg (50 mg to 100 mg for East Asians) and further from 200 mg to 300 mg once daily (100 mg to 150 mg for East Asians) based on the platelet response and safety data after two weeks of current dose level. After all participants finished the 8 week treatment period, platelet response and safety were analyzed before initiating Part 2 of the study. Supportive standard of care was allowed as needed. The duration of Part 1 was 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Part 1: Eltrombopag | Part 2: Placebo | Part 2: Eltrombopag | Total
Number analyzed (Participants) | 17 | 47 | 98 | 162
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.5 (10.78) | 70.6 (10.72) | 72.3 (8.94) | 71.8 (9.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 16 | 32 | 55
  Male | 10 | 31 | 66 | 107
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 0 | 0 | 1 | 1
  Asian - East Asian Heritage | 3 | 5 | 9 | 17
  Asian - South East Asian Heritage | 0 | 2 | 2 | 4
  White - Arabic/North African Heritage | 0 | 1 | 5 | 6
  White - White/Caucasian/European Heritage | 14 | 39 | 81 | 134

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Platelet Response up to Week 8 During Part 1
Description: A participant was considered as a responder if he/she met the following response criteria: a Baseline platelet count <20 Giga cells per liter (Gi/L) and a post-Baseline increased to >20 Gi/L and at least 2 times the Baseline value; or a Baseline platelet count >=20 Gi/L and a post-Baseline absolute platelet count increased to >=50 Gi/L and at least 2 times the Baseline value. The response criteria was evaluated at each visit. Increase in platelet count observed up to 3 days after a platelet transfusion was not considered as a platelet response. The Part 1 Population was comprised of all participants enrolled into Part 1.
Time Frame: From Baseline up to Week 8 during Part 1
Population: Part 1 Population: all subjects who enrolled in Part 1.
Measure: Number; unit: Participants
Arm/Group | Part 1: Eltrombopag
Number analyzed (Participants) | 17
Participants | 4

2. Primary Outcome: Clinically Relevant Thrombocytopenic Events (CRTE) From Week 5 up to Week 12 During Part 2
Description: A participant was considered to have a CRTE at a given assessment if he/she had platelet counts <10 Gi/L, or platelet transfusions, or >=Grade 3 hemorrhagic adverse events. CRTEs during Weeks 5 to 12 were compared between treatments using a generalized linear mixed model. Average of weekly proportion of subjects with CRTE during Week 5 to 12 was estimated for each treatment. Intent to Treat (ITT) Population was comprised of all randomized participants during Part 2.
Time Frame: From Week 5 up to Week 12 during Part 2
Population: Part 2 Population (Intent-To-Treat (ITT) Population: all randomized subjects in part 2)
Measure: Mean (95% Confidence Interval); unit: percentages of participants
Arm/Group | Part 2: Placebo | Part 2: Eltrombopag
Number analyzed (Participants) | 47 | 98
percentages of participants | 69 [57 to 80] | 54 [43 to 64]
Statistical Analysis 1: Comparison: Part 2: Placebo vs Part 2: Eltrombopag; Test type: Superiority or Other; p = 0.0315, Generalized Linear Mixed Models; Odds Ratio (OR) = 0.202, 95% CI 2-sided [0.047 to 0.868]

3. Secondary Outcome: Plasma Eltrombopag Pharmacokinetic Concentration-Time Data - by Visit (Part 1 Subjects)
Time Frame: Day 1 to week 8
Population: Pharmacokinetic population: all subjects in All Subjects Population who had a PK blood sample obtained/analyzed.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Part 1: Eltrombopag
Number analyzed (Participants) | 17
ug/mL
  Baseline/day 1 (Pre-dose PK) | 0 (0)
  Day8 week 1 (Pre-dose PK) | 7.7 (3.96)
  Day15 week 2 (Pre-dose PK) | 7.2 (5.17)
  Day22 week 3 (Pre-dose PK) | 14.3 (10.63)
  Day29 week 3 (2-6hrs post-dose PK) | 20.8 (14.98)
  Day36 week 5 (Pre-dose PK) | 20.2 (16.37)
  Day43 week6 (2-6hrs post-dose PK) | 41.2 (32.56)
  Day50 week 7 (Pre-dose PK) | 30.4 (27.95)
  Day57 week 8 (2-6hrs post-dose PK) | 30.1 (18.99)

4. Secondary Outcome: Plasma Eltrombopag Pharmacokinetic Concentration-Time Data - by Visit (Part 2 Subjects)
Time Frame: Day 1 to week 12
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: ug/mL
Groups:
- Part 2: Eltrombopag: The eltrombopag starting dose the participants received was 100 mg daily (50 mg for participants of East Asian heritage). The dose of eltrombopag was escalated from 100 mg to 200 mg (50 mg to 100 mg for East Asians) and further from 200 mg to 300 mg once daily (100 mg to 150 mg for East Asians) based on the platelet response and safety data after two weeks of current dose level. After all participants finished the 8 week treatment period, platelet response and safety were analyzed before initiating Part 2 of the study. Supportive standard of care was allowed as needed. The duration of Part 1 was 8 weeks.
Arm/Group | Part 2: Eltrombopag
Number analyzed (Participants) | 97
ug/mL
  Baseline/day 1 (Pre-dose PK) | 0 (0)
  Day15 week 2 (Pre-dose PK) | 10.1 (5.54)
  Day22 week 3 (2-6hrs post-dose PK) | 24.0 (14.6)
  Day29 week 4 (Pre-dose PK) | 20.2 (13.61)
  Day43 week 6 (Pre-dose PK) | 29.0 (18.13)
  Day50 week 7 (2-6hrs post-dose PK) | 42.9 (22.37)
  Day57 week8 (Pre-dose PK) | 36.3 (20.91)
  Day71 week 10 (Pre-dose PK) | 33.5 (20.40)
  Day78 week 11 (2-6hrs post-dose PK) | 41.2 (24.91)
  Day85 week12 (Pre-dose PK) | 30.7 (18.03)

5. Secondary Outcome: Mean Number of Platelet Transfusions
Time Frame: Weeks 5 to 12
Population: Part 2 Population (Intent-to-Treat population)
Measure: Mean (Standard Deviation); unit: Number of platelet transfusions
Groups:
- Part 2: Eltrombopag: Part 2: Eltrombopag The eltrombopag starting dose the participants received was 100 mg daily (50 mg for participants of East Asian heritage). The duration of treatment with the initial dose level prior to first dose escalation was determined based on the platelet response and toxicity observed in Part 1. The dose of eltrombopag was escalated from 100 mg to 200 mg (50 mg to 100 mg for East Asians) and further from 200 mg to 300 mg once daily (100 mg to 150 mg for East Asians) based on the platelet response and safety data after two weeks of current dose level. Supportive standard of care was allowed as needed throughout the study.
Arm/Group | Part 2: Eltrombopag | Part 2: Placebo
Number analyzed (Participants) | 98 | 47
Number of platelet transfusions | 18.8 (18.60) | 15.7 (20.36)

6. Secondary Outcome: Hematologic Improvement
Description: Definitions of hematologic improvement for platelets, neutrophils, and hemoglobin were based on modified International Working Group (IWG) consensus criteria.
Time Frame: Weeks 5 to 12
Population: Part 2 Population (Intent-to-Treat population)
Measure: Number; unit: Number of subjects
Arm/Group | Part 2: Eltrombopag | Part 2: Placebo
Number analyzed (Participants) | 98 | 47
Number of subjects
  Any Improvement | 10 | 4
  Platelets | 8 | 2
  Neutrophils | 4 | 4
  Hemoglobin | 0 | 0
  Platelets and neutrophils | 2 | 2
  Platelets and hemoglobin | 0 | 0
  Platelets, hemoglobin and neutrophils | 0 | 0
  Neutrophils and hemoglobin | 0 | 0

7. Secondary Outcome: Change in Mean Platelet Count
Time Frame: Baseline to Week 12
Population: Part 2 Population (Intent-to-Treat population)
Measure: Mean (Standard Deviation); unit: Gi/L
Arm/Group | Part 2: Eltrombopag | Part 2: Placebo
Number analyzed (Participants) | 98 | 47
Gi/L
  Day8 week1 | 3.36 (11.795) | 1.66 (6.249)
  Day15 week2 | 10.41 (60.225) | 3.06 (9.675)
  Day22 week3 | 6.23 (22.872) | 2.13 (9.258)
  Day29 week4 | 5.63 (17.582) | 2.44 (11.215)
  Day36 week5 | 8.58 (22.504) | 5.9 (16.000)
  Day43 week6 | 8.64 (19.779) | 5.93 (21.960)
  Day50 week7 | 9.91 (25.561) | 6.74 (31.074)
  Day57 week8 | 9.67 (23.243) | 7.84 (34.213)
  Day64 week9 | 12.84 (27.272) | 6.75 (31.709)
  Day71 week10 | 15.97 (33.866) | 6.23 (30.941)
  Day78 week11 | 14.42 (36.901) | 6.92 (26.906)
  Day 85 week12 | 9.06 (28.259) | 4.85 (26.219)

8. Secondary Outcome: Maximum Duration of Platelet Transfusion Independence
Time Frame: Weeks 5 to 12
Population: Part 2 Population (Intent-to-Treat population)
Measure: Mean (Standard Deviation); unit: maximum duration of platelet transfusion
Arm/Group | Part 2: Eltrombopag | Part 2: Placebo
Number analyzed (Participants) | 98 | 47
maximum duration of platelet transfusion | 26.3 (21.47) | 25.4 (19.70)

9. Secondary Outcome: Number of Participants With Maximum Bleeding Grade According to World Health Organization on Bleeding Scale
Description: Occurrence and severity of bleeding, measured using the WHO Bleeding Scale Grade 0=no bleeding; Grade 1=petechiae; Grade 2=mild blood loss; Grade 3=gross blood loss; Grade 4=debilitating blood loss.
Time Frame: Weeks 5 to 12
Population: Part 2 Population (Intent-to-Treat population)
Measure: Number; unit: Number of subjects
Arm/Group | Part 2: Eltrombopag | Part 2: Placebo
Number analyzed (Participants) | 98 | 47
Number of subjects
  Grade 0 (no bleeding) | 15 | 4
  Grade 1 (petechiae) | 31 | 22
  Grade 2 (mild blood loss) | 41 | 14
  Grade 3 (gross blood loss) | 5 | 3
  Grade 4 (debilitating blood loss) | 1 | 3
  Grades 0 - 1 | 46 | 26
  Grades 1 - 4 | 78 | 42
  Grades 2 - 4 | 47 | 20

10. Secondary Outcome: Independent Reviewer-Assessed Best Response
Description: Participants were evaluated in accordance with the modified International Working Group (Cheson, 2006). CR: Bone marrow blasts <5%, Hgb ≥11g/dL, Hematologic Improvement - Platelets (Baseline <20Gi/L: >20 Gi/L and 2x baseline; Baseline ≥20 Gi/L: ≥50 Gi/L and 2x baseline), Neutrophils ≥1.0 Gi/L, Peripheral blasts 0%. PR: Bone marrow blasts decreased by ≥50% but >5%, Peripheral blood as in CR. Marrow CR: Bone marrow blasts <5% and decrease by ≥50%, Note any Hematologic Improvements, Stable disease: Failure to achieve PR, but no evidence of progression for >8w, Cytogenetic response: Complete: disappearance of chromosomal abnormality; no new abnormalities Partial: ≥50% reduction of chromosomal abnormality.
Time Frame: up to week 12
Population: Part 2 Population (Intent-to-Treat population)
Measure: Number; unit: Number of subjects
Arm/Group | Part 2: Eltrombopag | Part 2: Placebo
Number analyzed (Participants) | 98 | 47
Number of subjects
  Responder | 1 | 1
  Complete response (CR) | 0 | 0
  Morphologic CR | 0 | 1
  Morphologic leukemia-free state | 0 | 0
  Marrow CR | 1 | 0
  Cytogenetic CR | 0 | 0
  Molecular CR | 0 | 0
  Non-responder | 97 | 46
  Partial response | 0 | 0
  Stable disease (non-responder) | 18 | 10
  Progressive disease (non-responder) | 41 | 28
  Not evaluable (non-responder) | 36 | 8
  Missing (non-responder) | 2 | 0

11. Secondary Outcome: Independent Reviewer Assessed Disease Progression
Time Frame: Up to week 12
Population: Part 2 Population (Intent-to-Treat population)
Measure: Number; unit: Number of subjects
Arm/Group | Part 2: Eltrombopag | Part 2: Placebo
Number analyzed (Participants) | 98 | 47
Number of subjects
  Disease progression | 61 (21.47) | 36 (19.70)
  No disease progression | 12 | 6
  Not evaluable | 23 | 5
  Missing | 2 | 0

12. Secondary Outcome: Median Overall Survival
Time Frame: Up to 13 months
Population: Part 2 Population (Intent-to-Treat population)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2: Eltrombopag | Part 2: Placebo
Number analyzed (Participants) | 98 | 47
Months | 4.27 [2.96 to 7.59] | 4.6 [3.29 to 7.82]

13. Secondary Outcome: Summary of Health Outcomes
Description: The number of subject with medical resource utilization (MRU) data are reported in this table.
  MRU included number of emergency room visits, number of home healthcare visits, number of hospitalization days, number of medication or surgery specialist visits, number of procedures inpatient, number of procedures outpatient, number of non-study radiology visits, number of non-study laboratory visits, number of nurse practitioner/physician assistance/nurse visits, number of primary care physician visits, number of telephone consultations.
Time Frame: week 12
Population: Part 2 Population (Intent-to-Treat population)
Measure: Number; unit: Subject with Events
Arm/Group | Part 2: Eltrombopag | Part 2: Placebo
Number analyzed (Participants) | 98 | 47
Subject with Events
  Number of emergency room visits (n=17, n=10) | 1 | 0
  Number of home healthcare visits (n=17, n=10) | 2 | 1
  Number of hospitalization days (n=17, n=10) | 5 | 4
  Number of med/surg specialist visits (n=17, n=10) | 1 | 3
  Number of procedures inpatient (n=17, n=10) | 2 | 1
  Number of procedures outpatient (n=17, n=10) | 1 | 1
  Number of non-study radiology visits (n=2, n=2) | 2 | 2
  Number of nurse prac/pa/nurse visits (n=17, n=10) | 5 | 3
  Number of primary care physician visits (n=17,10) | 7 | 1
  Number of telephone consultations (n=17, n=10) | 1 | 0
  Number of non-study laboratory visits (n=17, n=10) | 8 | 6

14. Secondary Outcome: Functional Assessment of Cancer Therapy (FACT)
Description: The FACT-Th-18 is the most widely used and accepted tool evaluating health-related quality-of-life outcomes in cancer patients with chronically low platelets (where Th designates thrombocytopenia). The entire FACT-Th-18 was used in this trial, which includes the 18-item thrombocytopenia subscale used to assess the impact of symptoms, signs, and functional consequences of thrombocytopenia in MDS and AML subjects. The FACT-Th-18 is a validated and reliable instrument with known psychometric properties. FACT-ThS is an 18 item questionnaire specific to assessing the impact of symptoms, signs, and functional consequences of Thrombocytopenia. ThS score ranges from 0 to 72 with higher the score, the better the QoL. FACT G total score moves from 0 to 108 where higher the score, the better the HRQL.
  FACT-Th Total Score is calculated by adding the FACT-ThS and FACT-G score. Total score ranges from 0 to 180 and again, higher the score, the better the HRQL.
Time Frame: Change from baseline, up to week 12
Population: Part 2 Population (Intent-to-Treat population)
Measure: Mean (Standard Error); unit: Adjusted mean change from baseline
Arm/Group | Part 2: Eltrombopag | Part 2: Placebo
Number analyzed (Participants) | 98 | 47
Adjusted mean change from baseline
  FACTG week 5 (n=61. n=34) | -0.79 (1.64) | -3.15 (2.19)
  FACTG week 9 (n=46. n=28) | -4.83 (1.82) | -2.76 (2.34)
  FACTG week12 (n=37. n=26) | -3.38 (1.94) | -4.17 (2.39)
  FACTHTOI week 5 (n=61, n=34) | 0.91 (2.04) | -2.28 (2.74)
  FACTHTOI week 9 (n=46, n=28) | -1.69 (2.24) | 0.19 (2.89)
  FACTHTOI week 12 (n=37, n=26) | -0.26 (2.37) | -1.56 (2.95)

15. Secondary Outcome: EQ-5D Utility Score Analysis
Description: EuroQoL Five Dimensions Questionnaire (EQ-5D) is a standardized generic preference based health related quality of life instrument. It records how one's health is "today" and consists of a descriptive system. The Descriptive system is Comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each dimension on the EQ-5D involves a 3-point response scale which indicates the level of impairment (level 1 = no problem; level 2 = some or moderate problem(s) and level 3 = unable, or extreme problems). Level of problem reported in each EQ-5D dimension determines a unique health state which is converted into a weighted health state index by applying scores from EQ-5D preference weights elicited from general population samples. This generates a unique description of the subjects' health status, which is valued between 0 (representing death) and 1 (representing perfect health). Higher the score, the better the quality of life.
  EQ-ED is a score.
Time Frame: Change from baseline, up to week 12
Population: Part 2 Population (Intent-to-Treat population)
Measure: Mean (Standard Error); unit: Adjusted mean change from baseline
Arm/Group | Part 2: Eltrombopag | Part 2: Placebo
Number analyzed (Participants) | 98 | 47
Adjusted mean change from baseline
  Week 5 (n=55. n=34) | -0.01 (0.04) | -0.15 (0.05)
  Week 9 (n=43. n=27) | -0.08 (0.04) | -0.06 (0.05)
  Week 12 (n=36. n=26) | -0.09 (0.05) | -0.11 (0.05)

ADVERSE EVENTS:
Groups:
- Eltrombopag, Part 1 Subjects: Eltrombopag, Part 1 subjects
- Eltrombopag, Part 2 Plus 1 Day From Part 2 Subjects: Eltrombopag, Part 2 plus 1 day from Part 2 subjects
- Placebo, Part 2 Plus 1 Day From Part 2 Subjects: Placebo, Part 2 plus 1 day from Part 2 subjects
- Eltrombopag, Part 3 Plus 30 Days From Part 2 Subjects: Eltrombopag, Part 3 plus 30 Days from Part 2 subjects
Arm/Group | Eltrombopag, Part 1 Subjects | Eltrombopag, Part 2 Plus 1 Day From Part 2 Subjects | Placebo, Part 2 Plus 1 Day From Part 2 Subjects | Eltrombopag, Part 3 Plus 30 Days From Part 2 Subjects
Serious Adverse Events (participants affected / at risk) | 9/17 | 56/97 | 32/47 | 39/59
Other Adverse Events (participants affected / at risk) | 17/17 | 89/97 | 44/47 | 54/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag, Part 1 Subjects (N=17) | Eltrombopag, Part 2 Plus 1 Day From Part 2 Subjects (N=97) | Placebo, Part 2 Plus 1 Day From Part 2 Subjects (N=47) | Eltrombopag, Part 3 Plus 30 Days From Part 2 Subjects (N=59)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 7 | 7 | 6
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Splenic artery thrombosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1 | 1 | 3
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Adrenal disorder (Endocrine disorders) | 0 | 0 | 0 | 1
Retinal vein occlusion (Eye disorders) | 0 | 1 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 3 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 2
Chest discomfort (General disorders) | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 1 | 0
Disease progression (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 1
General physical health deterioration (General disorders) | 0 | 2 | 2 | 2
Malaise (General disorders) | 0 | 0 | 0 | 1
Multi-organ failure (General disorders) | 0 | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 2 | 0
Pyrexia (General disorders) | 2 | 7 | 6 | 7
Sudden death (General disorders) | 0 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Abscess neck (Infections and infestations) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 4
Catheter site cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0 | 0
Cholecystitis infective (Infections and infestations) | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1
Endocarditis (Infections and infestations) | 0 | 0 | 0 | 1
Enteritis infectious (Infections and infestations) | 0 | 0 | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 2 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 1
Lung infection (Infections and infestations) | 0 | 1 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 14 | 5 | 10
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Sepsis (Infections and infestations) | 4 | 8 | 5 | 6
Septic shock (Infections and infestations) | 2 | 1 | 1 | 3
Splenic abscess (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 1
Streptococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 3 | 1 | 5
Urosepsis (Infections and infestations) | 0 | 1 | 1 | 0
Viral oesophagitis (Infections and infestations) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 1
International normalised ratio increased (Investigations) | 0 | 1 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 1 | 1
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 1
Syncope (Nervous system disorders) | 0 | 2 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1
Arterial thrombosis (Vascular disorders) | 0 | 1 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag, Part 1 Subjects (N=17) | Eltrombopag, Part 2 Plus 1 Day From Part 2 Subjects (N=97) | Placebo, Part 2 Plus 1 Day From Part 2 Subjects (N=47) | Eltrombopag, Part 3 Plus 30 Days From Part 2 Subjects (N=59)
Anaemia (Blood and lymphatic system disorders) | 3 | 8 | 2 | 2
Blood disorder (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 4 | 0 | 2
Haemolysis (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 3 | 1 | 4
Neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 2 | 3
Pericardial effusion (Cardiac disorders) | 1 | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 2 | 2
Conjunctival haemorrhage (Eye disorders) | 1 | 2 | 4 | 0
Eye haemorrhage (Eye disorders) | 0 | 5 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 1 | 0 | 0
Ocular icterus (Eye disorders) | 0 | 0 | 0 | 5
Abdominal pain (Gastrointestinal disorders) | 1 | 6 | 3 | 5
Abdominal pain upper (Gastrointestinal disorders) | 0 | 6 | 2 | 2
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 12 | 0 | 7
Diarrhoea (Gastrointestinal disorders) | 4 | 20 | 5 | 11
Gingival bleeding (Gastrointestinal disorders) | 1 | 13 | 8 | 7
Gingival swelling (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 9 | 7 | 7
Nausea (Gastrointestinal disorders) | 1 | 13 | 8 | 14
Vomiting (Gastrointestinal disorders) | 2 | 6 | 5 | 6
Asthenia (General disorders) | 3 | 4 | 5 | 6
Catheter site related reaction (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 23 | 3 | 9
Oedema peripheral (General disorders) | 0 | 9 | 3 | 7
Pain (General disorders) | 1 | 2 | 1 | 2
Pyrexia (General disorders) | 4 | 18 | 10 | 12
Xerosis (General disorders) | 1 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 3 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Arthritis infective (Infections and infestations) | 1 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 3 | 2
Escherichia infection (Infections and infestations) | 1 | 0 | 1 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 7
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 3 | 1 | 2
Skin infection (Infections and infestations) | 1 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 2 | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 5 | 2 | 3
Contusion (Injury, poisoning and procedural complications) | 1 | 4 | 3 | 5
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 3
Laceration (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 2 | 3 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 10 | 5 | 5
Aspartate aminotransferase increased (Investigations) | 1 | 3 | 5 | 2
Blood albumin decreased (Investigations) | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 2 | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 6 | 2 | 5
Blood phosphorus decreased (Investigations) | 1 | 0 | 0 | 0
Blood sodium increased (Investigations) | 1 | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 2 | 3 | 2
Body temperature fluctuation (Investigations) | 1 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 1 | 0
Platelet count decreased (Investigations) | 1 | 1 | 0 | 1
Serum ferritin increased (Investigations) | 2 | 1 | 0 | 1
Weight decreased (Investigations) | 1 | 1 | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 2 | 14 | 7 | 10
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 1 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 7 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 4 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 9 | 3 | 8
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 5 | 0 | 3
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 11 | 4 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 6 | 5 | 2
Aphonia (Nervous system disorders) | 1 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 9 | 4 | 2
Headache (Nervous system disorders) | 3 | 3 | 3 | 1
Mental impairment (Nervous system disorders) | 1 | 0 | 0 | 1
Poor quality sleep (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 2 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 2 | 0 | 2
Confusional state (Psychiatric disorders) | 0 | 1 | 1 | 3
Initial insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Azotaemia (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 2 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 13 | 4 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 9 | 5 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 27 | 11 | 12
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 3 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Blood blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 3
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 7 | 6 | 6
Petechiae (Skin and subcutaneous tissue disorders) | 6 | 41 | 11 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 1
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 3
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 2 | 3 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 7 | 9 | 9
Haemorrhage (Vascular disorders) | 2 | 4 | 4 | 1
Hypertension (Vascular disorders) | 0 | 6 | 0 | 0
Hypotension (Vascular disorders) | 1 | 3 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.